CLINICAL TRIAL: NCT04038008
Title: Single Dose Crossover Comparative Bioavailability Study of Fluconazole 200 mg Tablets Versus Diflucan® 200 mg Hard Capsules in Healthy Adult Subjects Under Fasting Conditions
Brief Title: Single Dose Crossover Comparative Bioavailability Study of Two Formulations of Fluconazole 200 mg in Healthy Adult Subjects Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmtechnology LLC (Industry)
Collaborators: Altasciences Company Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: PTL-P3-438 (v. 1.0 2019/07/12)
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Bioequivalence
Keywords: fluconazole; Diflucan®; bioequivalence
MeSH Terms: interventions — Fluconazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The randomization code will not be available to the personnel of the bioanalytical facility until the bioanalytical tables have been finalized and audited by the Quality Assurance (QA) department.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence AB (Other): 13 subjects assigned to the sequence AB will receive a single 200 mg dose of test product Fluconazole (1 x 200 mg tablet), marked as A in the sequence, in Period 1 and a single 200 mg dose of reference product Diflucan® (1 x 200 mg hard capsule), marked as B in the sequence, in period 2. These treatments will be administered orally with approximately 240 mL of water at ambient temperature, in the morning, following a minimum of 10-hour overnight fast. The tablet or hard capsule must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Fluconazole; Drug: Diflucan®
- Sequence BA (Other): 13 subjects assigned to the sequence BA will receive a single 200 mg dose of reference product Diflucan® (1 x 200 mg hard capsule), marked as B in the sequence, in Period 1 and test product Fluconazole (1 x 200 mg tablet), marked as A in the sequence, in Period 2. These treatments will be administered orally with approximately 240 mL of water at ambient temperature, in the morning, following a minimum of 10-hour overnight fast. The tablet or hard capsule must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Fluconazole; Drug: Diflucan®

INTERVENTIONS:
Drug: Fluconazole — Fluconazole is manufactured by Pharmtechnology LLC, Republic of Belarus. Each tablet contains 200 mg of fluconazole.
  Other Names: Test Product
Drug: Diflucan® — Diflucan® is manufactured by Fareva Amboise, France (MAH: PFIZER PHARMA PFE GmbH, Germany). Each hard capsule contains 200 mg of fluconazole.
  Other Names: Reference Product

SUMMARY:
This single dose study is designed in accordance with EMA (the European Medicines Agency) regulatory guidelines, with the aim of characterizing the comparative bioavailability of fluconazole in the two formulations in healthy subjects. As this is a bioequivalence trial where each subject will receive each study treatment in a crossover fashion, a control group is not included. Within the clinical portion of the study each subject will receive a single oral dose of the test and the reference formulation in compliance with the generated randomization code. The primary study endpoints are the pharmacokinetic (PK) parameters Cmax and AUC0-t of fluconazole.

DETAILED DESCRIPTION:
This is a single center, randomized, 2-treatment, 2-period, 2-sequence, crossover, single dose study design, in which 26 healthy adult subjects will receive one of the study treatments during each study period.

The objective of this study is to determine the bioequivalence of two different formulations of fluconazole after a single oral dose administration under fasting conditions. The secondary objective of this study is to determine the safety and tolerability of the Test product compared to the Reference formulation in healthy subjects.

Subject eligibility for this study will be determined at the screening visit and eligible subjects will be admitted to the clinical research unit at least 10 hours prior to drug administration for each study period.

A subject who withdraws or is withdrawn during the pretrial evaluations but before receiving the IP will not be considered as a drop-out and will not be included in the final database. Standbys should be recruited and available to replace any subject who withdraws prior to the first drug administration. On-study drop-outs will not be replaced.

Altasciences will generate the randomization code with a computer program according to the study design, the number of subjects and the sequence of treatment administration. The random allocation of each sequence of treatment administration to each subject will be done in such a way that the study is balanced. Once generated, the randomization code will be final and will not be modified.

For each study period, subjects will receive a single 40 mg oral dose of olmesartan medoxomil (the test or the reference formulation). Study participants will be aware they will receive different formulations of the same drug, without being informed which product (Test or Reference) is being administered.The date and time of each dose will be recorded. For each subject, all scheduled postdose activities and assessments will be performed relative to the time of study drug administration.

Subjects will fast overnight (no food or drink except water), for a minimum of 10 hours prior to dosing. Fasting will continue for at least 4 hours following drug administration, after which a standardized lunch will be served. A supper and a light snack will be served at appropriate times thereafter, but not before 9 hours after dosing.

A total of 22 blood samples will be collected (one tube of 4 mL each) in each study period for PK assessments. The first blood sample will be collected prior to drug administration while the others will be collected up to 120 hours after drug administration.

The analyte to be measured in the present study will be fluconazole. Fluconazole plasma concentrations will be measured according to a validated bioanalytical method.

Subjects are to be discharged from the clinic after the 24-hour postdose PK sample collection, and following medical approval. However, they may be advised to stay at the clinical site for safety reasons, if judged necessary by the physician in charge. Subjects will return to the clinic for blood collections at 48, 72, 96, and 120 hours postdose.

The expected terminal elimination half-life of fluconazole is 34 hours. To avoid any carry-over effect, a wash-out of 21 calendar days is planned between drug administrations.

The decision of which subjects will be included in the PK analysis is to be documented by the pharmacokineticist (or delegate) and approved by the sponsor before the start of the sample analysis by the bioanalytical facility. Subjects who are expected to provide evaluable PK data for both the Test and Reference products (based on viable PK samples) will be included in the PK analysis. Concentration data of the remaining subjects will be presented separately. Subjects who do not complete the sampling schedule of one or more study periods may be included in the PK and statistical analysis and bioequivalence determination for only the PK parameters that are judged not to be affected by the missing sample(s).

The parameter Tmax will be analyzed using a non-parametric approach. Test of fixed period, sequence and treatment effects will be based on the Wilcoxon's rank sum test (Mann-Whitney U-test). When appropriate (e.g. small or sparse sample), the exact version of the test will also be presented. All primary endpoints will be statistically analyzed using an ANOVA model. The fixed factors included in this model will be the subject effect (nested within sequence), the treatment received, the period at which it was given, as well as the sequence in which each treatment is received.

The treatment, sequence and period effects will the evaluated at the 5% significance level. Explanations for significant effects will be provided for log transformed PK parameters.

The 90% confidence interval for the exponential of the difference in LSmeans between the Test and Reference product will be calculated for the ln-transformed parameters (Test to Reference ratio of geometric LSmeans).

Statistical inference of fluconazole will be based on a bioequivalence approach using the following standards:

1. The ratio of geometric LSmeans with corresponding 90% confidence interval calculated from the exponential of the difference between the Test and Reference for the lntransformed parameters Cmax and AUC0-T should all be within the 80.00 to 125.00% bioequivalence range.
2. In case if AUC0-T is less than 80% of AUC0-∞ in more than 20% of the observations, truncated AUC0-72 will be used for bioequivalence assessment instead of AUC0-T. The ratio of geometric LSmeans with corresponding 90% confidence interval calculated from the exponential of the difference between the Test and Reference for the ln-transformed parameters Cmax and AUC0-72 should all be within the 80.00 to 125.00% bioequivalence range.

The safety population will include all subjects who received at least one formulation (Test or Reference). Safety assessments will include physical examination, clinical laboratory test and AE monitoring. Additional safety measurements may be performed at the discretion of the investigator for reasons related to subject safety.

Total study duration: up to 55 days (including screening).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (ICF)
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Healthy Caucasian adult male or female
4. If female, meets one of the following criteria:

   1. Is of childbearing potential and agrees to use one of the accepted contraceptive regimens from at least 28 days prior to the first study drug administration through to at least 30 days after the last dose of the study drug. An acceptable method of contraception includes one of the following:

      * Abstinence from heterosexual intercourse
      * Systemic contraceptives (combined birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch)
      * Intrauterine device (with or without hormones)
      * Male condom with spermicide or male condom with a vaginal spermicide (gel, foam, or suppository)
      * Male partner vasectomized at least 6 months prior to the first study drug administration

      Or
   2. Male partner has had a vasectomy less than 6 months prior to dosing, and agrees to use an additional acceptable contraceptive method from the first study drug administration through to at least 30 days after the last dose of the study drug

      Or
   3. Is of non-childbearing potential, defined as surgically sterile (i.e. has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or is in a postmenopausal state (i.e. at least 1 year without menses without an alternative medical condition prior to the first study drug administration)
5. Aged at least 18 years but not older than 55 years
6. Body mass index (BMI) within 18.5 kg/m2 to 30.0 kg/m2, inclusively
7. Non- or ex-smoker (An ex-smoker is defined as someone who completely stopped using nicotine products for at least 180 days prior to the first study drug administration)
8. Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without clinical significance, as determined by an investigator
9. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination (including vital signs) and/or ECG, as determined by an investigator

Exclusion Criteria:

1. Female who is lactating at screening
2. Female who is pregnant according to the pregnancy test at screening or prior to the first study drug administration
3. History of significant hypersensitivity to fluconazole, any related azole compounds, or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
4. Presence or history of significant gastrointestinal, liver or kidney disease, or any other condition that is known to interfere with drug absorption, distribution, metabolism or excretion, or known to potentiate or predispose to undesired effects
5. History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
6. Presence of clinically significant ECG abnormalities at the screening visit, as defined by medical judgment
7. Seated blood pressure below 110/60 mmHg at the screening visit
8. History of rare hereditary problems of galactose and/or lactose intolerance, lactase deficiency or glucose-galactose malabsorption
9. Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
10. Any clinically significant illness in the 28 days prior to the first study drug administration
11. Use of any prescription drugs (with the exception of hormonal contraceptives or hormone replacement therapy) in the 28 days prior to the first study drug administration, that in the opinion of an investigator would put into question the status of the participant as healthy
12. Any history of tuberculosis
13. Positive test result for alcohol and/or drugs of abuse at screening or prior to the first drug administration
14. Positive screening results to HIV Ag/Ab Combo, Hepatitis B surface Antigen (HBsAG (B) (hepatitis B)) or Hepatitis C Virus (HCV (C)) tests
15. Inclusion in a previous group for this clinical study
16. Intake of fluconazole in the 28 days prior to the first study drug administration
17. Use of terfenadine, astemizole, erythromycin, quinidine, pimozide, or cisapride in the 7 days prior to the first study drug administration
18. Intake of an Investigational Product (IP) in the 28 days prior to the first study drug administration
19. Donation of 50 mL or more of blood in the 28 days prior to the first study drug administration
20. Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the 56 days prior to the first study drug administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) of fluconazole in plasma after administration of the test and the reference products | 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 12.00, 24.00, 48.00, 72.00, 96.00, 120.00 hours after each drug administration
  Maximum observed concentration in plasma
AUC0-T of fluconazole in plasma after administration of the test and the reference products | 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 12.00, 24.00, 48.00, 72.00, 96.00, 120.00 hours after each drug administration
  Cumulative area under the concentration time curve calculated from 0 to TLQC using the linear trapezoidal method, where TLQC represents time of last observed quantifiable concentration
AUC0-72 of fluconazole in plasma after administration of the test and the reference products (in case if AUC0-T is less than 80% of AUC0-∞ in more than 20% of the observations, truncated AUC0-72 will be used as primary endpoint instead of AUC0-T) | 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 12.00, 24.00, 48.00, 72.00, 96.00, 120.00 hours after each drug administration
  Cumulative area under the concentration time curve calculated from 0 to 72 hours using the linear trapezoidal method. Nominal time will be used to estimate AUC0-72 using the NCA built-in tool in Phoenix® WinNonlin®. Any actual time that deviates by more than 1 minute from the 72-hour time point will be extrapolated/intrapolated as per Phoenix® WinNonlin®'s built-in formulas.

SECONDARY OUTCOMES:
Tmax of fluconazole in plasma after administration of the test and the reference products | 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 12.00, 24.00, 48.00, 72.00, 96.00, 120.00 hours after each drug administration
  Time of maximum observed concentration; if it occurs at more than one time point, Tmax is defined as the first time point with this value
TLQC of fluconazole in plasma after administration of the test and the reference products | 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 12.00, 24.00, 48.00, 72.00, 96.00, 120.00 hours after each drug administration
  Time of last observed quantifiable concentration
AUC0-∞ of fluconazole in plasma after administration of the test and the reference products | 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 12.00, 24.00, 48.00, 72.00, 96.00, 120.00 hours after each drug administration
  Area under the concentration time curve extrapolated to infinity, calculated as AUC0-t + ĈLQC (the predicted concentration at time TLQC) / λZ (apparent elimination rate constant)
Residual area of fluconazole in plasma after administration of the test and the reference products | 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 12.00, 24.00, 48.00, 72.00, 96.00, 120.00 hours after each drug administration
  Extrapolated area (i.e. percentage of AUC0-INF due to extrapolation from TLQC to infinity)
Time point where the log-linear elimination phase begins (TLIN) of fluconazole in plasma after administration of the test and the reference products | 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 12.00, 24.00, 48.00, 72.00, 96.00, 120.00 hours after each drug administration
  Time point where the log-linear elimination phase begins
λZ of fluconazole in plasma after administration of the test and the reference products | 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 12.00, 24.00, 48.00, 72.00, 96.00, 120.00 hours after each drug administration
  Apparent elimination rate constant, estimated by linear regression of the terminal linear portion of the log concentration versus time curve
Terminal elimination half-life (Thalf) of fluconazole in plasma after administration of the test and the reference products | 0.00 (prior to each drug administration) and 0.17, 0.33, 0.50, 0.75, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 12.00, 24.00, 48.00, 72.00, 96.00, 120.00 hours after each drug administration
  Terminal elimination half-life, calculated as ln(2)/λZ
Number of treatment-emergent adverse events for the test and the reference products | Up to 30 days (after the first drug administration until 3 days following the last blood sample of the study)
  The safety population will include all subjects who received at least one dose of the test or the reference product. Any significant changes will be recorded as treatment-emergent adverse events only if they are judged clinically significant by the qualified investigator or delegate.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, MD, Principal Investigator — Altasciences Company Inc.
Locations (1):
- Altasciences Company Inc., Mount Royal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No